CLINICAL TRIAL: NCT01553942
Title: Afatinib Sequenced With Concurrent Chemotherapy and Radiation in EGFR-Mutant Non-Small Cell Lung Tumors: The ASCENT Trial
Brief Title: Afatinib With CT and RT for EGFR-Mutant NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lecia V. Sequist, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-464
Record Dates: First submitted 2012-03-05; First posted 2012-03-14 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Lung Neoplasms | interventions — Afatinib; Radiation; Cisplatin; Pemetrexed; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Afatinib (Experimental): Afatinib
  Interventions: Drug: Afatinib; Radiation: Radiation; Drug: Cisplatin; Drug: Pemetrexed; Procedure: Surgery

INTERVENTIONS:
Drug: Afatinib — induction phase-two 4 week cycles. consolidation phase-twenty six 4 week cycles
Radiation: Radiation — Daily, Monday-Friday
Drug: Cisplatin — Day 1 of each cycle, IV infusion over 60 minutes
Drug: Pemetrexed — Day 1 of each cycle, given as IV infusion over 10 minutes after cisplatin infusion
Procedure: Surgery — Surgery to remove tumor

SUMMARY:
This research study is a Phase II clinical trial. Phase II clinical trials test the effectiveness of an investigational drug to learn whether the drug works in treating a specific cancer. "Investigational" means that the drug is still being studied and that study doctors are trying to find out more about it-such as the safest dose to use, the side effects it may cause, and if the drug is effective for treating different types of cancer. It also means that the FDA has not yet approved the drug for the patients type of cancer or for any use outside of research studies.

Chemotherapy and radiation is the standard treatment for the patients with stage III non-small cell lung cancer (NSCLC). For people with epidermal growth factor receptor (EGFR) mutations, adding a type of drug called a tyrosine kinase inhibitor (TKI) can help increase the response to treatment.

Afatinib is a tyrosine kinase inhibitor. It has been studied in a previous research study in participants with more advanced NSCLC. Results from that study indicate it may be helpful in treating NSCLC with EGFR mutations.

In this study, patients with stage III NSCLC and EGFR mutations will receive the standard treatment of radiation and chemotherapy. If possible, the patients tumor will be removed by surgery. Afatinib will be given before radiation and chemotherapy and after surgery. The aim of giving afatinib before radiation therapy is to try to shrink the tumor. This may make the radiation therapy more effective since radiation therapy tends to work better on smaller tumors.

The goal of this study is to see if adding afatinib to standard treatment helps to improve the response to treatment.

DETAILED DESCRIPTION:
Study treatment will be divided into 5 stages:

Stage 1-induction, consisting of afatinib for two 4-week cycles. Afatinib is a pill that the patient takes by mouth once per day. The patient will receive a study drug diary in which to record the doses of afatinib.

Stage 2-concurrent radiation and chemotherapy with cisplatin/pemetrexed for two 3-week cycles.

Stage 3-Surgery to remove tumor for participants whose tumor can be removed by surgery. This will be done about 4-6 weeks after finishing radiation and chemotherapy. The exact timing will depend upon how quickly the patient recovers from side effects of the radiation and chemotherapy. The investigators will use a piece of the patients tumor removed by surgery for research tests to look for biomarkers such as genes and proteins that may be associated with response to afatinib, chemotherapy or radiation.

Stage 4-Chemotherapy after surgery (adjuvant chemotherapy). The patients doctor will decide if the patient will receive chemotherapy after the patients surgery but before receiving consolidation with afatinib. If the patient does receive this, it will start 6-12 weeks after surgery or finishing radiation if the patient does not have surgery. The chemotherapy will be the same as that received along with the radiation therapy.

Stage 5-Consolidation with afatinib for twenty-six 4-week cycles (2 years) for participants who responded to the 2 cycles of induction afatinib.

The investigators would like to keep track of the patients medical condition and status of the patients disease for up to 5 years after the patient stops study treatment. Keeping in touch with the patients and checking on the patients condition every year helps the investigators look at the long-term effects of the research study. The patients will be asked to have CT scans as follows:

* Every 3 months for the first year after stopping study treatment
* Every 6 months for years 2-4 after stopping study treatment
* Once per year in year 5 after stopping study treatment

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IIIA NSCLC
* Measurable disease
* Have lung cancer harboring an EGFR mutation
* Must be evaluated by a medical oncologist, radiation oncologist and thoracic surgeon within 4 weeks of enrollment into study to document that they are a candidate for chemoradiation and for consideration of surgical resection (not required to be a surgical candidate)

Exclusion Criteria:

* Pregnant or breastfeeding
* Prior EGFR TKI therapy
* Prior treatment with radiation to the thoracic region (including breast irradiation)
* Known pre-existing interstitial lung disease
* Significant or recent gastrointestinal disorders with diarrhea as a major symptom
* History or presence of relevant cardiovascular abnormalities
* Any other concomitant serious illness or organ system dysfunction
* Active hepatitis B, C or known HIV carrier
* Known or suspected active drug or alcohol use
* Known hypersensitivity to afatinib, cisplatin, or pemetrexed
* Concomitant treatment with strong inhibitor of P-gp
* History of an active malignancy within the last 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 2 years
  Assess the response rate to induction afatinib.

SECONDARY OUTCOMES:
2 Year Progression-Free Survival | 2 years
  Estimate the 2-year progression-free survival (PFS)
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 years
  Describe the number of patients that have side effects of various types from the study treatment
Unresectable Disease Converted to Operable Cases | 2 years
  Estimate the proportion of patients with initially unresectable disease that can be converted to operable cases
Locoregional Tumor Control Rates | 2 years
  Estimate 2-year locoregional tumor control rates, distant metastasis rates and overall survival rates, as well as median overall survival (OS)
Evaluation of EGFR Mutation Status and other genotypes | 2 years
  Evaluate the status of various relevant genes such as EGFR, MET, and other genes that might be related to response or resistance to afatinib, and assess relationship to clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Lecia V Sequist, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts